CLINICAL TRIAL: NCT00631657
Title: A 6-Month, Double-Blind, Randomized, Placebo-Controlled, Parallel Group Outpatient Trial, Investigating the Efficacy and Safety of Org 50081 in Adult Patients With Chronic Primary Insomnia
Brief Title: A 6-Month Efficacy and Safety Study of Org 50081 in Adult Patients With Chronic Primary Insomnia (21106/P05701/MK-8265-002)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P05701; 21106 (Other: Organon Protocol Number); 2007-005236-92 (EudraCT Number)
Record Dates: First submitted 2008-02-29; First posted 2008-03-10 (Estimated); Results first posted 2014-08-01 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Sleep Initiation and Maintenance Disorders; Mental Disorders; Dyssomnias; Sleep Disorders; Sleep Disorder, Intrinsic
Keywords: placebo controlled; randomized; double blind
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Mental Disorders; Dyssomnias; Sleep Wake Disorders; Sleep Disorders, Intrinsic | interventions — Mirtazapine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Esmirtazapine 4.5 mg (Experimental): Participants receive esmirtazapine 4.5 mg tablets, administered once a day for 6 months
  Interventions: Drug: Esmirtazapine
- Placebo (Placebo Comparator): Participants receive placebo tablets, administered once a day for 6 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Esmirtazapine — One esmirtazapine 4.5 mg tablet once a day
  Arms: Esmirtazapine 4.5 mg
Drug: Placebo — One placebo tablet once a day
  Arms: Placebo

SUMMARY:
To investigate the long-term efficacy and safety of treatment with esmirtazapine (Org 50081, SCH 900265, MK-8265) compared to placebo, in participants with chronic primary insomnia. Primary efficacy variable is Total Sleep Time (TST).

DETAILED DESCRIPTION:
Insomnia is a common complaint or disorder throughout the world. About one third of the population in the industrial countries reports difficulty initiating or maintaining sleep, resulting in a non-refreshing or non-restorative sleep. The majority of the insomniacs suffer chronically from their complaints.

The maleic acid salt of Org 4420, code name Org 50081 (esmirtazapine), was selected for development in the treatment of insomnia. The first clinical trial with esmirtazapine was a proof-of-concept trial with a four-way cross-over design. All 3 esmirtazapine dose groups showed a statistically significant positive effect on TST (objective and subjective) and Wake Time After Sleep Onset (WASO), as compared to placebo.

The current study is designed to assess the long-term efficacy and safety of esmirtazapine in a double-blind, randomized, placebo-controlled, parallel group outpatient trial in participants suffering from chronic primary insomnia. During the 6-month treatment period, participants are randomly assigned to receive either esmirtazapine or placebo. Then, during the 7-day discontinuation period, participants who received esmirtazapine in the 6-month treatment period are randomly assigned to receive either esmirtazapine or placebo, while participants who received placebo in the 6-month treatment period continue to receive placebo.

ELIGIBILITY:
Inclusion Criteria:

* are at least 18 and less than 65 years;
* sign written informed consent after the scope and nature of the investigation have been explained;
* have shown capability to complete the LogPad questionnaires;
* have difficulty falling asleep, maintaining sleep or have early morning awakening;

Exclusion Criteria:

* Significant medical or psychiatric illness causing sleep disturbances.
* Have a history of bipolar disorder or attempted suicide or have a family (immediate family) history of suicide.
* Have a sleep disorder such as sleep-related breathing disorder, restless leg syndrome, narcolepsy.
* Significant other medical illness such as acute or chronic pain, heart-, kidney-, or liver disease within the last year.
* Currently diagnosed or meet the criteria for Major Depressive Disorder (MDD) or have been treated for MDD in the last 2 years.
* Substance abuse, excessive use of alcohol (determined by the physician) or drug addiction within the last year.
* Are night workers or rotating shift workers or plan to travel through more than 3 time-zones.
* Routinely nap during the day.
* Have a Body Mass Index (BMI) of 36 or more.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Actual)
Dates: Start 2008-03-04 (Actual); Primary Completion 2009-11-19 (Actual); Study Completion 2009-11-19 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Ivgy-May N, Hajak G, van Osta G, Braat S, Chang Q, Roth T. Efficacy and safety of esmirtazapine in adult outpatients with chronic primary insomnia: a randomized, double-blind placebo-controlled study and open-label extension. J Clin Sleep Med. 2020 Sep 15;16(9):1455-1467. doi: 10.5664/jcsm.8526. PMID 32351205

RESULTS

PARTICIPANT FLOW:
Groups:
- Esmirtazapine 4.5 mg/Esmirtazapine 4.5 mg: Participants receive esmirtazapine 4.5 mg tablets, administered once a day (QD) for 6 months, then participants receive esmirtazapine 4.5 mg tablets, administered QD for 7 days
- Esmirtazapine 4.5 mg/Placebo: Participants receive esmirtazapine 4.5 mg tablets, administered QD for 6 months, then participants receive placebo tablets, administered QD for 7 days
- Placebo/Placebo: Participants receive placebo tablets, administered QD for 6 months, then participants receive placebo tablets, administered QD for 7 days
Period: 6-Month Treatment Period
Arm/Group | Esmirtazapine 4.5 mg/Esmirtazapine 4.5 mg | Esmirtazapine 4.5 mg/Placebo | Placebo/Placebo
Started | 344 | 0 | 116
Treated | 342 (Two randomized participants were not treated during the 6-month Treatment Period.) | 0 | 115 (One randomized participant was not treated during the 6-month Treatment Period.)
Completed | 203 | 0 | 66
Not Completed | 141 | 0 | 50
Not completed — Adverse Event | 47 | 0 | 7
Not completed — Withdrawal by Subject | 14 | 0 | 5
Not completed — Lack of Efficacy | 34 | 0 | 25
Not completed — Lost to Follow-up | 7 | 0 | 2
Not completed — Uncooperative Reasons Unrelated to Trial | 21 | 0 | 6
Not completed — Other | 16 | 0 | 4
Not completed — Not Treated | 2 | 0 | 1
Period: 7-Day Discontinuation Period
Arm/Group | Esmirtazapine 4.5 mg/Esmirtazapine 4.5 mg | Esmirtazapine 4.5 mg/Placebo | Placebo/Placebo
Started | 67 (One participant was radomized in the Discont. Period, without completing the Treatment Period.) | 137 | 66
Treated | 66 (One participant was not treated during the Discontinuation Period.) | 136 (One participant was not treated during the Discontinuation Period.) | 65 (One participant was not treated during the Discontinuation Period.)
Completed | 65 | 136 | 65
Not Completed | 2 | 1 | 1
Not completed — Not Treated | 1 | 1 | 1
Not completed — Other | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Baseline Analysis Population consists of all participants who received study drug. Two participants in the esmertazapine 4.5 mg group and one participant in the placebo group did not receive study drug.
Groups:
- Esmirtazapine 4.5 mg: Participants receive esmirtazapine 4.5 mg tablets, administered QD for 6 months
- Placebo: Participants receive placebo tablets, administered QD for 6 months
- Total: Total of all reporting groups
Arm/Group | Esmirtazapine 4.5 mg | Placebo | Total
Number analyzed (Participants) | 342 | 115 | 457
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.4 (11.4) | 49.0 (11.1) | 47.8 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 210 | 71 | 281
  Male | 132 | 44 | 176

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total Sleep Time (TST) - 6-Month Treatment Period
Description: TST was defined as the time recorded for sleep diary question 6 "How much time did you actually spend sleeping?" as reported by participants using a LogPad (hand-held electronic data capture device). Baseline was defined as the mean TST from the Placebo Run-in Period. Change from Baseline was calculated as the mean of combined data from Weeks 14 through 26, using a last observation carried forward (LOCF) approach.
Time Frame: Baseline and the Mean of Weeks 14-26
Population: The Intent-To-Treat (ITT) population consisted of all participants who received at least one dose of study drug and had a baseline and at least one postbaseline TST efficacy assessment.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Esmirtazapine 4.5 mg | Placebo
Number analyzed (Participants) | 342 | 115
minutes | 65.9 (71.9) | 19.3 (62.1)
Statistical Analysis 1: Comparison: Esmirtazapine 4.5 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Difference in Least Squares (LS) Means = 48.7, 95% CI 2-sided [35.0 to 62.5] — ANCOVA performed with fixed effects for treatment and (pooled) center as factors and baseline TST as covariate

2. Secondary Outcome: Number of Participants Who Experienced Adverse Events (AEs)
Description: An AE is defined as any unfavorable and unintended change in the structure, function or chemistry of the body whether or not considered related to study drug. The number of participants who experienced AEs is combined for the 6-Month Treatment Period and the 7-Day Discontinuation Period.
Time Frame: Up to 31 weeks
Population: The All-Subjects-Treated (AST) population consisted of all participants who received at least one dose of any study drug.
Measure: Number; unit: participants
Groups:
- Placebo: Participants receive placebo tablets, administered QD
Arm/Group | Esmirtazapine 4.5 mg | Placebo
Number analyzed (Participants) | 342 | 115
participants | 253 | 75

3. Secondary Outcome: Number of Participants Who Discontinued Study Drug Due to an AE
Description: An AE is defined as any unfavorable and unintended change in the structure, function or chemistry of the body whether or not considered related to study drug. The number of participants who discontinued study drug due to an AE is combined for the 6-Month Treatment Period and the 7-Day Discontinuation Period.
Time Frame: Up to 27 weeks
Population: The AST population consisted of all participants who received at least one dose of any study drug.
Measure: Number; unit: participants
Arm/Group | Esmirtazapine 4.5 mg | Placebo
Number analyzed (Participants) | 342 | 115
participants | 47 | 7

4. Secondary Outcome: Change From Baseline in Sleep Latency (SL) - 6-Month Treatment Period
Description: SL was defined as the time recorded for sleep diary question 3 "How long did it take you to fall asllep?", as reported by participants using a LogPad. Baseline was defined as the mean SL from the Placebo Run-in Period. Change from Baseline was calculated as the mean of combined data from Weeks 14 through 26, using an LOCF approach.
Time Frame: Baseline and the Mean of Weeks 14-26
Population: The ITT population consisted of all participants who received at least one dose of study drug and had a baseline and at least one postbaseline SL efficacy assessment.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Esmirtazapine 4.5 mg | Placebo
Number analyzed (Participants) | 342 | 115
minutes | -29.7 (47.3) | -26.9 (46.8)
Statistical Analysis 1: Comparison: Esmirtazapine 4.5 mg vs Placebo; Test type: Superiority or Other; p = 0.2145, ANCOVA; Difference in LS Means = -4.9, 95% CI 2-sided [-12.6 to 2.8] — ANCOVA performed with fixed effects for treatment and (pooled) center as factors and baseline SL as covariate

5. Secondary Outcome: Change From Baseline in Wake Time After Sleep Onset (WASO) - 6-Month Treatment Period
Description: WASO was defined as the time recorded for sleep diary question 5 "How much time were you awake, after falling asleep initially?", as reported by participants using a LogPad. Baseline was defined as the mean WASO from the Placebo Run-in Period. Change from Baseline was calculated as the mean of combined data from Weeks 14 through 26, using an LOCF approach.
Time Frame: Baseline and the Mean of Weeks 14-26
Population: The ITT population consisted of all participants who received at least one dose of study drug and had a baseline and at least one postbaseline WASO efficacy assessment.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Esmirtazapine 4.5 mg | Placebo
Number analyzed (Participants) | 342 | 115
minutes | -46.4 (57.7) | -20.8 (51.4)
Statistical Analysis 1: Comparison: Esmirtazapine 4.5 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Difference in LS Means = -25.0, 95% CI 2-sided [-34.5 to -15.4] — ANCOVA performed with fixed effects for treatment and (pooled) center as factors and baseline WASO as covariate

6. Other Pre Specified Outcome: Change From Baseline in Number of Awakenings (NAW) - 6-Month Treatment Period
Description: NAW was defined as the number of times recorded for sleep diary question 4a "How many times did you wake up during the night?", as reported by participants using a LogPad. Baseline was defined as the mean NAW from the Placebo Run-in Period. Change from Baseline was calculated as the mean of combined data from Weeks 14 through 26, using an LOCF approach.
Time Frame: Baseline and the Mean of Weeks 14-26
Population: The ITT population consisted of all participants who received at least one dose of study drug and had a baseline and at least one postbaseline NAW efficacy assessment.
Measure: Mean (Standard Deviation); unit: number of awakenings
Arm/Group | Esmirtazapine 4.5 mg | Placebo
Number analyzed (Participants) | 342 | 115
number of awakenings | -0.8 (1.2) | -0.5 (0.9)

7. Other Pre Specified Outcome: Change From Baseline in Sleep Quality - 6-Month Treatment Period
Description: Sleep Quality was assessed using a Visual Analog Scale (VAS) in response to the sleep diary question 7 "Rate the quality of your sleep last night", as reported by participants using a LogPad. Responses could range from 0=Very poor to 100=Excellent, with a higher score indicating greater sleep quality. Baseline was defined as the mean Sleep Quality score from the Placebo Run-in Period. Change from Baseline was calculated as the mean of combined data from Weeks 14 through 26, using an LOCF approach.
Time Frame: Baseline and the Mean of Weeks 14-26
Population: The ITT population consisted of all participants who received at least one dose of study drug and had a baseline and at least one postbaseline Sleep Quality efficacy assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Esmirtazapine 4.5 mg | Placebo
Number analyzed (Participants) | 342 | 115
score on a scale | 16.1 (19.5) | 5.8 (14.0)

8. Other Pre Specified Outcome: Change From Baseline in Satisfaction With Sleep Duration - 6-Month Treatment Period
Description: Satifaction with Sleep Duration was assessed using a Visual Analog Scale (VAS) in response to the sleep diary question 8 "How satisfied are you about your sleep duration of last night?", as reported by participants using a LogPad. Responses could range from 0=Very unsatisfied to 100=Fully satisfied, with a higher score indicating great satisfaction with sleep duration. Baseline was defined as the mean Satisfaction with Sleep Duration score from the Placebo Run-in Period. Change from Baseline was calculated as the mean of combined data from Weeks 14 through 26, using an LOCF approach.
Time Frame: Baseline and the Mean of Weeks 14-26
Population: The ITT population consisted of all participants who received at least one dose of study drug and had a baseline and at least one postbaseline Satisfaction with Sleep Duration efficacy assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Esmirtazapine 4.5 mg | Placebo
Number analyzed (Participants) | 342 | 115
score on a scale | 18.3 (20.1) | 7.2 (15.9)

9. Other Pre Specified Outcome: Change From Baseline in Two Aggregate Measures of Short Form 36 (SF-36) Health Survey Score - 6-Month Treatment Period
Description: SF-36 is a participant-rated questionnaire that consists of 8 scaled scores: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each of the 8 questions carries equal weight. The SF-36 can be divided into 2 aggregate summary measures: the Physical Component Summary (PCS) and the Mental Component Summary (MCS). The scores can range from 0 to 100, with a lower score indicating more disability. Baseline was defined as the SF-36 score assessed at randomization.
Time Frame: Baseline and Week 26
Population: The ITT population consisted of all participants who received at least one dose of study drug and had a baseline and a Week 26 SF-36 efficacy assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Esmirtazapine 4.5 mg | Placebo
Number analyzed (Participants) | 189 | 63
score on a scale
  Change from BL at Week 26 - PCS | 1.6 (6.8) | -0.2 (6.0)
  Change from BL at Week 26 - MCS | 4.6 (10.8) | 4.5 (9.1)

10. Other Pre Specified Outcome: Change From Baseline in Investigator Global Rating (IGR) - 6-Month Treatment Period
Description: The IGR is a clinician-rated 7-point scale used to assess the severity of illness. Severity is rated on a scale from 1=Normal to 7=Extremely severe. Baseline was defined as the last non-missing value obtained during the Placebo Run-in Period. IGR assessments were done at Baseline of the 6-Month Treatment Period and and at the end of the 6-Month Treatment Period to assess the effects of treatment.
Time Frame: Baseline and Week 26
Population: The ITT population consisted of all participants who received at least one dose of study drug and had a baseline and a Week 26 IGR efficacy assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Esmirtazapine 4.5 mg | Placebo
Number analyzed (Participants) | 200 | 65
score on a scale | -2.1 (1.4) | -1.4 (1.4)

11. Other Pre Specified Outcome: Change From Baseline in Investigator Global Rating (IGR) - 7-Day Discontinuation Period
Description: The IGR is a clinician-rated 7-point scale used to assess the severity of illness. Severity is rated on a scale from 1=Normal to 7=Extremely severe. Baseline was defined as the last non-missing value obtained during the Placebo Run-in Period. IGR assessments were done at Baseline of the 6-Month Treatment Period and and at the end of the 7-day Discontinuation Period to assess the effects of discontinuing treatment.
Time Frame: Baseline and End of 7-day Discontinuation Period
Population: The ITT population consisted of all participants who received at least one dose of study drug and had a baseline and a 7-Day Discontinuation Period IGR efficacy assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Esmirtazapine 4.5 mg/Esmirtazapine 4.5 mg: Participants receive esmirtazapine 4.5 mg tablets, administered QD for 6 months during the Treatment Period, followed by esmirtazapine 4.5 mg tablets, administered QD for 7 days during the Discontinuation Period
- Esmirtazapine 4.5 mg/Placebo: Participants receive esmirtazapine 4.5 mg tablets, administered QD for 6 months during the Treatment Period, followed by placebo tablets, administered QD for 7 days during the Discontinuation Period
- Placebo/Placebo: Participants receive placebo tablets, administered QD for 6 months during the Treatment Period, followed by placebo tablets, administered QD for 7 days during the Discontinuation Period
Arm/Group | Esmirtazapine 4.5 mg/Esmirtazapine 4.5 mg | Esmirtazapine 4.5 mg/Placebo | Placebo/Placebo
Number analyzed (Participants) | 59 | 128 | 60
score on a scale | 0.3 (0.7) | 0.5 (1.0) | 0.0 (0.7)

ADVERSE EVENTS:
Time Frame: Up to 30 days after last dose of study drug (up to 31 weeks)
Description: AE data include AEs that occurred during the 6-month Treatment Period and the 7-day Discontinuation Period. AEs are reported for the study drug participants were receiving at the time the AE occurred.
Groups:
- Esmirtazapine 4.5 mg: Participants receive esmirtazapine 4.5 mg tablets, administered QD
Arm/Group | Esmirtazapine 4.5 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 8/342 | 2/115
Other Adverse Events (participants affected / at risk) | 183/342 | 40/115
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Esmirtazapine 4.5 mg (N=342) | Placebo (N=115)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Retinal vein occlusion (Eye disorders) | 1 (1) | 0 (0)
Sudden visual loss (Eye disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Infectious mononucleosis (Infections and infestations) | 1 (1) | 0 (0)
Cartilage injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Synovial rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nerve compression (Nervous system disorders) | 1 (1) | 0 (0)
Bunion operation (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Esmirtazapine 4.5 mg (N=342) | Placebo (N=115)
Dry mouth (Gastrointestinal disorders) | 20 (21) | 5 (5)
Fatigue (General disorders) | 18 (20) | 7 (7)
Nasopharyngitis (Infections and infestations) | 35 (42) | 14 (17)
Weight increased (Investigations) | 58 (63) | 4 (4)
Increased appetite (Metabolism and nutrition disorders) | 34 (37) | 1 (1)
Dizziness (Nervous system disorders) | 27 (29) | 4 (4)
Headache (Nervous system disorders) | 30 (35) | 14 (21)
Somnolence (Nervous system disorders) | 51 (56) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less